CLINICAL TRIAL: NCT06567301
Title: Extracorporeal Shockwave Versus Phonophoresis on Functional and Anatomical Changes Detected With Artificial Intelligence Technology in Knee Osteoarthritis
Brief Title: Extracorporeal Shockwave Versus Phonophoresis Using Chitosan-Nanoparticles Gel on Functional and Anatomical Changes Detected With Artificial Intelligence Based Texture Analysis Algorithm in Knee Osteoarthritis Patients: A Double Blind Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Athar Tarek Mohamed Fahmy Azab, principle Investigators, Cairo University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: P.T.REC/012/005026
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Chitosan Nanoparticles Gel; Artificial Intelligence Texture Analysis Bases Algorithm; Subchondral Bone Changes (Anatomical Changes); Extracorporeal Shockwave
Keywords: knee osteoarthritis; chitosan nanoparticles gel; artificial intelligence; texture analysis; artificial intelligence texture analysis bases algorithm; chitosan; subchondral bone changes; anatomical changes; Extracorporeal shockwave; ultrasound therapy; Phonophoresis; medical imaging; knee OA pathogenesis; pathophysiology
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded controlled randomized study (pretest-posttest measurement)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Ultrasound therapy combined with Chitosan nanoparticles gel and Exercises Program (Experimental): In this group will receive ultrasound therapy coupled with chitosan-nanoparticles gel with an exercises program. The US protocol which will consist of pulsed ultrasound waves. The parameters that will be selected consists of; frequency of 1 MHz, 1 W/cm2 power delivered at an intensity of an intensity of 2.5W/ cm2 and with duty cycle of 25% and will be applied with a 5-cm diameter applicator.
  The area of treatment will be cleaned to permit an effective skin applicator coupling. Each patient will be placed in a supine position for the application of ultrasound. A suitable palpation to locate the discomfort source and some passive motions to identify a range of motion restriction will be completed prior to the ultrasound application.
  Ultrasound will be applied to the medial and lateral aspects of the knee in circular motions, with the probe at right angles to ensure maximum absorption of energy. Each session will last for 5 minutes.
  Interventions: Combination Product: Ultrasound therapy combined with Chitosan nanoparticles gel
- Group B: Application of Extracorporeal Shockwave and Exercises Program: (Active Comparator): This group will receive ESWT with an exercises program. Subjects will receive 5 sessions, one week apart. Before the treatment, subjects will be placed in supine to expose and prepare the treated area with the knee flexed at angle of 90° and the hip is abducted and externally rotated. The impulses will be applied on the subchondral bone at the medial and lateral tibia condyle at 2.0 cm below the joint line in anteroposterior view and 2.0 cm from the medial skin edge in lateral view. The treatment application will be as follows: 2000 impulses will be administered at (EFD) with an energy flux density ranging from 0.22-0.43 mJ / mm2 at 8 Hz. In which 0.22 mJ/mm²: likely corresponds to around 1.5-3 bars, while 0.43 mJ/mm² likely corresponds to around 3-5 bars. The probe was chosen effective treatment depth (5-20-mm focal depth), semi-movable technique of the shockwave applicator and 5 minutes duration.
  Interventions: Combination Product: Ultrasound therapy combined with Chitosan nanoparticles gel
- Group C: Exercises Program (Placebo Comparator): Patients in this group will receive only an exercises program for 3 times weekly for 4 weeks. This program includes:
  (1) Warming-up (5 min); (2) strengthening exercises for the lower limbs: 3 sets of 15 repetitions: flexion SLR, abduction SLR, and extension SLR, standing knee flexion, quadriceps isometrics, 10 repetitions of 5 s, 0° and 30°; (3) aerobic exercise on a stationary bike (20 min), (4) and stretching (5 min) with a weekend break.
  All patients in the three groups (A, B and C) will receive the same exercise program.
  Interventions: Combination Product: Ultrasound therapy combined with Chitosan nanoparticles gel

INTERVENTIONS:
Combination Product: Ultrasound therapy combined with Chitosan nanoparticles gel — Gymna - Belgian
  Other Names: Extracorporeal Shockwave Therapy

SUMMARY:
A parallel double blinded randomized controlled clinical trial (RCT) with a 1:1:1 allocation will be conducted in an orthopedic clinic in Cairo and Giza Governments - Egypt.

This RCT will evaluate the pain reduction, self-reported functional improvement, physical functional and anatomical improvement following the application of phonophoresis using chitosan-nanoparticles gel, ECSW therapy and traditional exercises compared to each other.

The treatment period will last for 4 weeks with a total of (12 sessions/ 3 sessions per week for the application of phonophoresis using chitosan-nanoparticles gel and traditional exercises program) and (5 sessions/ 1 every week for the application of ECSWT). The participants will be assessed at two different time-points (before-after treatment) with a sample size of 40 patients in each group (3 groups)

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common degenerative disease that is ranked as the 10th largest contributor to disabilities that has a link to higher comorbidity and excess mortality. One of most common degenerative diseases is knee osteoarthritis (KOA). KOA is a progressive, chronic degenerative condition that places a heavy socioeconomic burden on healthcare systems and society. The prevalence of knee OA has sharply increased to more than the double in the last 10 years as result of steady state in life expectancy.

KOA is a well-known as a cartilage disease that involves degradation and loss of articular cartilage. However, OA is usually accompanied by changes in the subchondral bone, with sclerosis, bone cyst, and osteophyte formation.

Recent studies reported that subchondral bone remodeling plays a very important role in KOA, mediating and preceding cartilage damage. The increase in subchondral bone stiffness decreases the ability to scatter the loading forces within the knee joint, which then increases the force loaded on articular cartilage. Therefore, the cartilage damage and progress of OA accelerated over time. The focus of treatment in early KOA have shifted from the articular cartilage to the subchondral bone and become a potential therapeutic target of various therapeutic methods.

Regarding KOA pain, accumulating evidence suggests that bottom-up vascularization from subchondral bone plays a larger role than top-down vessel invasion originating from synovial tissue or synovium during cartilage erosion in OA. As a result, it is a common complaint of orthopedists that osteoarthritis pain is not associated with the radiographic presentation. Recent work revealed a relatively weak relationship between cartilage loss and OA joint pain.

As different approaches aimed at articular cartilage or synovial components had inefficient results and the mechanism of bone cartilage crosstalk is gradually becoming clear, this study will try to confirm the critical role of subchondral bone in knee osteoarthritis and that subchondral bone could be an ideal outcome measure of osteoarthritis treatment.

Low-intensity pulsed ultrasound (LIPUS) and extracorporeal shockwave therapy (ECSWT) are effective as a non-invasive method in histopathological recovery with more intense sight, ECSWT has shown effectiveness in the regression of early KOA associated with improving the subchondral bone remodeling, decrease the number of osteophytes and it can also increase osteocytes activity. Besides, ECSWT could alleviate chronic inflammatory activities in the whole joint through down-regulating inflammatory cytokines. Additionally, it was reported that application of ESWT to the subchondral bone of the knee significantly increased bone volume and trabecular number and reduced bone porosity. Overall, ESWT could reverse the pathology of OA progression to some extent.

Low-intensity US might influence the subchondral bone unit under joint disuse. LIUS with its associated acoustic radiation force can alleviate subchondral bone sclerosis during OA progression under normal joint use. In addition, if US technology combined with bioactive compounds materials as chitosan (CS), could improve the encapsulation efficiency of bioactive compounds whereas not only reduced the nanoparticle size but also narrowed their size distribution, this makes US as an effective delivery of biomaterials such as chitosan. In this context, inclusion of mixed interventions with US could improve its effect. Therefore, this study will couple the use of US therapy with a new green environmentally friendly material called chitosan in the form of a topical gel.

Chitosan appears as proteoglycan in the extracellular matrix (shells) of some species of cephalopods. Chitosan's biocompatibility, gradual degradability, non-toxicity, biological activity, anti-inflammatory properties, and antibacterial action, makes chitosan regarded as the best material for hydrogel. Some studies used CS as intra-articular injection for KOA and concluded that CS can promote chondrocyte proliferation, block inflammatory and catabolic mediators. Therefore, Phonophoresis using chitosan could reduce inflammation, limit cartilage degeneration and improve subchondral bone remodeling process.

Additionally, it is well known that confirming diagnosis of KOA is based on assessing joint space width and this is carried out through radiography which depends on the Kellgren-Lawrence grade (K-LG) scale. Despite K-LG scale is considered the most used classical diagnostic tool for KO, it has several drawbacks, including its application to the progression of diseases, its insensitivity to change, or inconsistencies in the authors' initial descriptions. Furthermore, it is limited in how it evaluates treatment efficacy because it mostly uses pain scores.

By looking to the adverse effects of conventional radiology, many studies had reported the possibility of an allergic reaction, expensive costs, lengthy inspection times, and difficulties in scanning patients with specific conditions.

Taking this into account, artificial intelligence (AI)-based approaches are starting to be used to solve these issues as image identification, pre-operative risk assessment, clinical decision- making, and analysis of large data sets, diagnosis, monitor, prognosis of rheumatological diseases, identifying risk factors for complications and has the unique ability to anticipate outcomes using patient-specific algorithms. AI plays a vital role in the appraisal of treatment, in which key progress in the clinical practice of rheumatology is the innovation of advanced imaging modalities.

The use of AI in orthopedics has mostly concentrated on the development of Machine learning (ML) and deep learning (DL) on these pictures. Deep learning, which is a subset of ML, can assist in automatic interpretation of medical images, which may increase diagnostic accuracy and speed, flag the most urgent and critical patients for immediate attention, reduce the amount of human error caused by fatigue and/or inexperience, lessen the strain on medical professionals by reducing their workload, and, in general, improve orthopedic care.

Subchondral bone-remodeling process was reported previously as an important pathophysiology of KO whereas subchondral bone sclerosis is widely considered to be the hallmark of OA. Texture analysis (TA) algorithm is used to detect changes in the subchondral bone density during remodeling process. It was demonstrated encouraging findings and the potential of automated texture analysis employing an AI algorithm as a diagnostic tool for OA in comparison to traditional TA techniques. Bone structure value (BSV) is considered as a maximum-likelihood estimator of OA as automated TA depends on it in the analysis and assessment process that measures the micro-structure of the tibial subchondral bone depends on area of interest (ROI). Consequently, the purpose of this study is to explore the difference between ECSWT, LIUS and traditional exercises regarding the pain reduction, functional improvement (self-reported and physical function) and anatomical improvement of subchondral bone (trabecular tibial bone) micro-structural changes.

ELIGIBILITY:
Inclusion Criteria:

1. Age between ≥40 and ≤ 65 years old.
2. Both genders.
3. Patients should have OA of the knee, Kellgren-Lawrence scores of 2 and 3 on radiologic evaluation.
4. If both knees diagnosed as OA, the most affected one will be selected.
5. Diagnosis of KOA who had knee pain and functional disabilities for at least three months, according to American College of Rheumatology classification (ACR) at screening visit.
6. Visual Analogue Scale (VAS) at rest score of ≥40 mm.
7. Subjects have sufficient cognition that enables them to understand the requirements of the study, comply with the study procedures and visit schedule.

Exclusion Criteria:

1. Patients with any previous knee surgeries or lower limb fractures.
2. Chronic inflammatory diseases such as rheumatoid arthritis.
3. Any neurological disorders.
4. Moderate to significant knee synovitis.
5. Hot or red knee.
6. History and/or physical examination findings compatible with the internal derangement of knee.
7. Pregnancy.
8. Patients with BMI more than 35 (morbid obesity).
9. Absence of current physical therapy treatments for KOA.
10. Cognitive limitations or endocrine disease.
11. Patients who had undergone arthroscopy or treatment with intra-articular hyaluronic acid during previous 6 months.
12. Use of NSAIDs one week prior to screening visit.
13. Orthopedic diseases that may affect or interfere with the therapeutic effect.
14. Habitual use of psychotropic or narcotic analgesics for ≥1 week within 8 weeks prior to screening.
15. Participated in other intervention studies on the past 6 months to screening
16. Participants with congenital musculoskeletal deformity.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Anatomical improvement | one month
  subchondral bone improvement following the application of Phonophoresis using chitosan-nanoparticles gel, ECSW therapy and assessed by Artificial intelligence based texture analysis algorithm

SECONDARY OUTCOMES:
level of knee pain | one month
  by VAS

OTHER OUTCOMES:
Physical functional assessment | one month
  by TUG
Self-reported functional assessment | one month
  by the (ArWOMAC) Index for measurement of perceived health and physical function

CONTACTS AND LOCATIONS:
Overall Officials: Athar Tarek Mohamed Fahmy Azab, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Physical Therapy College - Cairo University, Giza, El Dokki
  - Physical therapy college - Cairo University, Giza, EL Doqqi